CLINICAL TRIAL: NCT01623570
Title: Prospective Randomized Open Label Study to Compare the Efficacy and Safety of Ovarian Stimulation With Pergoveris® and Menopur® in Women With Severe Luteinizing Hormone (LH) and Follicular Stimulating Hormone (FSH) Deficiency.
Brief Title: Clinical Outcomes in WHO Type I Anovulatory Women Using r-hFSH+r-hLH in a 2:1 Ratio or hMG-HP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Riproduzione e Andrologia (Other)
Responsible Party: Principal Investigator, Domenico Carone, MD, Centro Riproduzione e Andrologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREA022011
Record Dates: First submitted 2012-06-17; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: Luteinizing Hormone; Hypogonadotropic Hypogonadism; Ovulation Induction; Chorionic Gonadotropin
MeSH Terms: conditions — Hypogonadism | interventions — pergoveris; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pergoveris: 150IU r-hFSH+ 75IU r-hLH (Experimental): This is a prospective randomized study using two in-label treatments for the patient disease: Pergoveris and Menopur. Pergoveris arms can be considered as experimental for the aim of the study, anyway it is standard routine practice for HH women.
  Interventions: Drug: Pergoveris: 150IU r-hFSH + 75IU r-hLH
- Menopur: hMG-HP (150IU) (Experimental): This is a prospective randomized study using two in-label treatments for the patient disease: Pergoveris and Menopur. Menopur can be considered as experimental for the aim of the study, anyway it is standard routine practice for HH women
  Interventions: Drug: Menopur: HMG-HP (150 IU)

INTERVENTIONS:
Drug: Pergoveris: 150IU r-hFSH + 75IU r-hLH — Fixed formulation of two recombinant gonadotropins
  Other Names: Pergoveris
  Arms: Pergoveris: 150IU r-hFSH+ 75IU r-hLH
Drug: Menopur: HMG-HP (150 IU) — Human Menopausal Gonadotropin is an urinary estract from menopausal women containing 150IU of FSH and 150 IU of LH-like activity (HCG)
  Other Names: Menopur
  Arms: Menopur: hMG-HP (150IU)

SUMMARY:
The aim of the study is to compare the efficacy and safety of r-hFSH+r-hLH in a 2:1 ratio with human Menopausal Gonadotropin Highly Purified (hMG-HP), in WHO type I anovulation, HH women.

This open-label monocentric, randomized comparative trial, to receive the two different standard clinical practice treatments:

* 1 vial of Pergoveris: (vial/powder 150 International unit (IU) r-hFSH+ 75IU r-hLH)
* 2 vials of Menopur: (vials/powder hMG 75IU).

Follicular development were monitored until the protocol hCG requirement is met and a single injection of hCG was administered.

Main Outcome Measures were follicular development i.e. follicle ≥ 17 millimeters (mm), pre-ovulatory E2 ≥ 400 picomole/Liter (pmol/L) and mid-luteal phase Progesterone (P4) ≥ 25 nanomole/Liter (nmol/L).

DETAILED DESCRIPTION:
World Health Organization (WHO) type I hypogonadotropic anovulation (hypogonadotropic hypogonadism, HH) is a rare alteration of the reproductive system with absent or decreased function of the gonads, caused by congenital, including genetic, or acquired reduced hypothalamic or pituitary activity. This results in abnormally low serum levels of Follicular Stimulation Hormone (FSH) and Luteinizing Hormone (LH) and negligible oestrogen (E2) activity.

The most convenient treatment is daily injections of exogenous gonadotropins that has been proven to be effective.

Patients lacking an effective hypothalamic-pituitary activity (WHO type I anovulation) do not produce sufficient threshold levels of endogenous LH, which is required to obtain optimal follicular development and steroidogenesis when treated with FSH alone. Therefore a combination therapy with adequate doses of both FSH and LH in an optimal ratio is required in order to restore fertility.

The LH activity could be produced by LH itself or by human Chorionic Gonadotropin (hCG) and the two gonadotropins are available to be used in the WHO type I patients in two different formulations both in indication for this type of patients. It would be worth of interest to assess if these two different formulations could elicit the same clinical outcomes in standard clinical practice or not.

The aim of the study is to compare the efficacy and safety of recombinant human FSH and recombinant human LH (r-hFSH+r-hLH) in a 2:1 ratio with human Menopausal Gonadotropin Highly Purified (hMG-HP), containing LH-like activity, in women with severe LH and FSH deficiency (WHO type I anovulation, HH).

All patients were diagnosed with HH according to a negative progesterone (P4) challenge test, serum LH<1.2 IU/L and FSH <5 IU/L, a transvaginal ultrasound showing a uterus with a midline echo, no ovarian tumor or cyst and ≤ 13 small follicles (mean diameter ≤ 10millimeters (mm)) on the largest section through each ovary, a Body Mass Index (BMI) between 18 and 32 Kilograms for square meters(Kg/m2), and no systemic diseases.

In this open-label monocentric, randomized comparative trial, patients was randomized in two arms in 1:1 ratio, to receive the two different standard clinical practice treatments:

* 1 vial of Pergoveris: (vial/powder 150 International Units (IU) r-hFSH+ 75IU r-hLH)stimulation day 1 until required hCG level is met. The dose can be adjusted at stimulation Day 6 according to subject ovarian response and standard clinical practice
* 2 vials of Menopur: (vial/powder hMG containing 75IU FSH + 75IU LH-like activity). stimulation day 1 until required hCG level is met. The dose can be adjusted at stimulation Day 6 according to subject ovarian response and standard clinical practice Follicular development were monitored according clinical practice by ultrasound (US) and/or estradiol (E2) levels, until the protocol hCG requirement is met (i.e., at least one follicle greater than or equal to 17 mm). After this, a single injection of hCG was administered in order to induce final oocyte maturation.

Main Outcome Measures were ovulation induction as measured by follicular development i.e. follicle ≥ 17 mm, pre-ovulatory E2 ≥ 400 picomole/Liter (pmol/L) and mid-luteal phase Progesterone ≥ 25 nanomole/Liter (nmol/L). Secondary efficacy endpoints included estradiol levels/follicle at mid-cycle, number of follicles at mid-cycle and pregnancy rate (PR).

Drug safety was assessed by monitoring adverse events and the incidence of local reactions after drug injection at local site. Ovarian hyperstimulation syndrome (OHSS) was assessed and recorded according to Golan classification According to this protocol, patients were initially treated for one cycle. If consenting, patients who did not become pregnant during the first cycle were treated for a further optional one or two series of cycles with the same criteria of randomization, i.e. maintaining the same treatment as the previous cycle.

ELIGIBILITY:
Inclusion Criteria:

* WHO Type I HH Women
* Serum LH <1.2 IU/L
* Serum FSH <5 IU/L
* Age 25-36 years
* No ovarian tumor
* No cyst
* ≤ 13 small follicles (mean diameter ≤ 10mm)
* BMI between 18 - 32 Kg/m2
* no systemic diseases

Exclusion Criteria:

-

Ages: 25 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
E2 in pmol/L | Day after the protocol hCG requirement is met (at least one follicle of 17mm is monitored by ultrasound)
  Evaluate the patients steroidogenesis
Number of Follicles > 17mm | last US day before hCG administration
  To evaluate the efficacy of the stimulation and maturity of follicles
P4 in nmol/L | Day after the protocol hCG requirement is met (at least one follicle of 17mm by US)
  Progesteron level to evaluate the endometrial receptivity

SECONDARY OUTCOMES:
Endometrial thickness | Day 5 and Day 10 of stimulation treatment
  Evaluation of endometrial development and receptivity
Total number of Follicles | Last US day before hCG administration
  To evaluate the overall efficacy of stimulation treatment, also including follicles < 17mm
Clinical Pregnancy rate | days 35-42 post hCG
  Evaluate the ratio between primary end points and final stimulation outcome
Occurence of any adverse events (early or late ovarian hyperstimulation syndrome) | Days 15-20 post hCG

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Riproduzione e Andrologia, Taranto, Italy, Italy

REFERENCES:
- [Derived] Carone D, Caropreso C, Vitti A, Chiappetta R. Efficacy of different gonadotropin combinations to support ovulation induction in WHO type I anovulation infertility: clinical evidences of human recombinant FSH/human recombinant LH in a 2:1 ratio and highly purified human menopausal gonadotropin stimulation protocols. J Endocrinol Invest. 2012 Dec;35(11):996-1002. doi: 10.3275/8657. Epub 2012 Oct 22. PMID 23095369